CLINICAL TRIAL: NCT04561765
Title: Innovation in the Treatment of Persistent Pain in Adults With Neurofibromatosis Type 1 (NF1): Implementation of the iCanCope Mobile Application- Clinical Trial
Brief Title: Innovation in the Treatment of Persistent Pain in Adults With NF1: Implementation of the iCanCope Mobile Application- Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Hospital for Sick Children (Other); Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2000029045
Record Dates: First submitted 2020-09-10; First posted 2020-09-24 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neurofibromatosis 1; Chronic Pain
MeSH Terms: conditions — Neurofibromatosis 1; Chronic Pain

STUDY DESIGN:
Intervention Model Description: A 1x3 pilot randomized control trial (RCT) (iCanCope-NF, iCanCope-NF +Contingency Management (CM), Control Group) will be conducted with adults with NF1 who suffer from pain.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iCanCope (Experimental): In this group, individuals will receive the iCanCope-NF program. The intervention will be delivered on a restricted password-protected mobile application. Participants will be encouraged to log onto the pain diary app (via automated alerts) once per day over the 8-week period to complete pain diary entries and develop and track their goals related to their pain, physical, social activities, sleep, as well as work through content based on their goals.
  Interventions: Device: iCanCope
- iCanCope+Contingency Management (Experimental): In addition to the iCanCope-NF activities outlined above, individuals will be rewarded with incentives (contingency management) such as points that are redeemable for prize-based gift card vouchers. Points will be accrued through access to new sections, daily check-ins, and engagement of the mobile application. Based on research, the total amount of money that can be earned by the patient over the course of the two months is 50 dollars USD.
  Interventions: Device: iCanCope+Contingency Management
- Control Group (No Intervention): The control group is designed to assess for potential effects on outcomes of time, attention, during the study. In addition to usual care, participants will be required to complete baseline and follow-up assessments similar to that of the intervention groups. They will be given that patient education, through preapproved flyers and information found from national websites regarding pain management, but no self-management strategies or opportunities for social support. They will not have access to the mobile application during the course of experiment; however, the control group will be offered the full iCanCope-NF program following the trial (T2) for a period of 2 months after the study is over.

INTERVENTIONS:
Device: iCanCope — The iCanCope mobile and web-based self-management program has been empirically evaluated for multiple painful diseases
  Arms: iCanCope
Device: iCanCope+Contingency Management — In addition to the iCanCope-NF activities outlined above, individuals will be rewarded with incentives (contingency management) such as points that are redeemable for prize-based gift card vouchers. Points will be accrued through access to new sections, daily check-ins, and engagement of the mobile application. Based on research, the total amount of money that can be earned by the patient over the course of the two months is 50 dollars USD.
  Arms: iCanCope+Contingency Management

SUMMARY:
To demonstrate the initial feasibility and determine preliminary impact on clinical outcomes of the iCanCope-NF program in a pilot RCT. If successful this pilot study will support conducting a larger randomized control trial (RCT). The primary research question is what is the feasibility of the iCanCope-NF program? The investigators define feasibility as (1) rates of accrual and dropout, daily log-ins, engagement, and outcome measures completed and (2) perceptions regarding intervention acceptability and satisfaction; and what are the levels of engagement. log-ins, with the intervention? The secondary questions are: (1) how does the iCanCope-NF program compare with the control condition in differences of pain and pain-related activity limitations, sleep functioning, emotional functioning (depression, anxiety), opioid usage, pain catastrophizing, self-efficacy, respondent burden (i.e. Physical Functioning, R, Vitality, Social Functioning, Role-Emotional, and Mental Health), and psychological flexibility immediately post-treatment (T2), (2) does the iCanCope-NF + CM increase the engagement of the iCanCope-NF program as compared to iCanCope-NF without CM, and do their corresponding levels of pain and pain-related activity decrease with CM?, and (3) do individuals with NF1 utilize the Mindfulness based alternative approaches (MBAA) to help reduce pain symptoms? The investigators hypothesize that by customizing and including MBAA to the program for adults with NF1, that individuals who engage regularly as seen through Analytics Platform for Evaluating Effective Engagement (APEEE) application, will acquire new sets of skills to facilitate pain management, while pain as reported with the Brief Pain Inventory will decrease.

ELIGIBILITY:
Inclusion Criteria:

* adults 18+
* able to read and understand English at 5th grade level
* permanently reside in the United States
* have pain interference aggregate scores of three or more in the last two weeks using the Brief Pain Inventory-Short Form (BPI-SF) scale

Exclusion Criteria:

* have an undiagnosed case of NF1
* have documented major co-occurring psychiatric disease
* have moderate to severe cognitive deficits
* have depression assessed using the Patient Health Questionnaire (PHQ-9) or anxiety assessed using the Generalized Anxiety Disorder scale (GAD-7) greater than or equal to the appropriate thresholds (10=mild major depression; 5=mild severe anxiety)

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Frank D Buono, PHD, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other investigator. Only non-PHI/IPD will be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- iCanCop+Contingency Management: In addition to the iCanCope-NF activities outlined above, individuals will be rewarded with incentives (contingency management) such as points that are redeemable for prize-based gift card vouchers. Points will be accrued through access to new sections, daily check-ins, and engagement of the mobile application. Based on research, the total amount of money that can be earned by the patient over the course of the two months is 50 dollars USD.
  iCanCope+Contingency Management: In addition to the iCanCope-NF activities outlined above, individuals will be rewarded with incentives (contingency management) such as points that are redeemable for prize-based gift card vouchers. Points will be accrued through access to new sections, daily check-ins, and engagement of the mobile application. Based on research, the total amount of money that can be earned by the patient over the course of the two months is 50 dollars USD.
Period: Overall Study
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Started | 40 | 42 | 40
Completed | 38 | 36 | 34
Not Completed | 2 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group | Total
Number analyzed (Participants) | 40 | 42 | 40 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.9) | 40.9 (13.2) | 45.6 (10.5) | 42.4 (12.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 27 | 30 | 28 | 85
  Male | 12 | 12 | 12 | 36
  Other | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan | 0 | 0 | 1 | 1
  Asian | 1 | 2 | 0 | 3
  Black or African American | 2 | 4 | 4 | 10
  Other | 3 | 3 | 3 | 9
  White | 34 | 33 | 32 | 99
Region of Enrollment [Number; unit: participants]
  United States | 40 | 42 | 40 | 122
Marital Status [Count of Participants; unit: Participants]
  Divorced | 3 | 3 | 3 | 9
  Married | 13 | 15 | 20 | 48
  Other | 0 | 1 | 0 | 1
  Seperated | 2 | 0 | 0 | 2
  Single | 20 | 22 | 17 | 59
  Widowed | 1 | 1 | 0 | 2
  MIssing | 1 | 0 | 0 | 1
Degree [Count of Participants; unit: Participants]
  Advanced | 4 | 4 | 5 | 13
  Associates | 9 | 8 | 3 | 20
  Bachelors | 10 | 13 | 9 | 32
  High School or GED | 10 | 7 | 11 | 28
  Some college | 6 | 7 | 8 | 21
  Technical schooling | 1 | 2 | 3 | 6
  Missing | 0 | 1 | 1 | 2
Age at Diagnosis [Mean (Standard Deviation); unit: years] — Population: one participant had missing data from each group
  years
    number analyzed (Participants) | 39 | 41 | 39 | 119
    (all) | 11.7 (13.1) | 10.3 (11.8) | 11.5 (12.2) | 11.2 (12.3)
Surgeries [Count of Participants; unit: Participants] — Population: Collected fom completers
  Participants
    0 | 7 | 5 | 6 | 18
    1 to 3 | 14 | 17 | 12 | 43
    4 to 6 | 5 | 3 | 6 | 14
    7 to 10 | 2 | 3 | 5 | 10
    11 or more | 10 | 8 | 5 | 23
    Unknown or missing | 2 | 6 | 6 | 14
Parents [Count of Participants; unit: Participants]
  Yes | 13 | 14 | 22 | 49
  No | 20 | 24 | 17 | 61
  Maybe | 7 | 4 | 1 | 12
Children [Count of Participants; unit: Participants]
  Yes | 11 | 10 | 13 | 34
  No | 9 | 11 | 10 | 30
  Maybe | 1 | 1 | 2 | 4
  Missing | 19 | 20 | 15 | 54

OUTCOME MEASURES:

1. Primary Outcome: Engagement Activity
Description: Average minutes per day logged on the mobile application will be evaluated between the two groups using the mobile application.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | iCanCope | iCanCope+Contingency Management
Number analyzed (Participants) | 38 | 36
minutes per day | 4.7 (3.9) | 8.1 (6.5)

2. Primary Outcome: Pain Severity
Description: A comparison within groups change of pain severity measured by the Brief Pain Inventory-Short Form. Respondents rate items on a 0-10 scale to indicate the pain severity and interference, and the total score is the mean of each subfactor. The higher the score indicates more severity and interference of pain.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale
  Intake (Baseline) | 4.743 (1.83) | 4.625 (2.17) | 4.787 (2.15)
  Discharge (about 2 weeks) | 4.164 (1.99) | 3.778 (2.48) | 4.875 (2.65)
  Follow-Up (on average 4 months) | 4.439 (2.01) | 4.160 (2.44) | 4.375 (2.47)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P values at discharge; Test type: Superiority; p = 0.051, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; P values at discharge; Test type: Superiority; p = 0.206, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; P values at discharge; Test type: Superiority; p = 0.765, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P values at follow-up; Test type: Superiority; p = 0.991, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; P values at discharge; Test type: Superiority; p = 0.963, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; P values at discharge; Test type: Superiority; p = 0.916, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

3. Primary Outcome: Pain Interference Index
Description: A comparison within groups change of pain interference measured by the Pain Interference Index Scale. Respondents rate items on a 0-6 scale to indicate how much pain has interfered with various activities, and the total score is the mean of the six items. Where 6 indicates high interference. Presented here are the non-linear converted T scores with a 'population' mean of 50 and standard deviation of 10. Scores above 50 indicate more pain interference.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
T-score
  Intake (Baseline) | 57.709 (8.68) | 58.666 (7.92) | 59.394 (7.41)
  Discharge (an average of 2 weeks) | 57.033 (7.45) | 54.965 (7.78) | 60.210 (9.21)
  Follow-Up (on average 4 months) | 57.783 (8.04) | 56.366 (9.47) | 59.424 (9.73)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P value at discharge; Test type: Superiority; p = 0.005, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; P value at discharge; Test type: Superiority; p = 0.270, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; P value at discharge; Test type: Superiority; p = 0.177, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P Value at follow-up; Test type: Superiority; p = 0.300, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; Test type: Superiority; p = 0.996, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; Test type: Superiority; p = 0.334, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

4. Secondary Outcome: Treatment Services Review
Description: What are perceptions of satisfaction across groups exposed to the iCanCope mobile application using an The Treatment Services Review (TSR). Data presented here represents the themes that emerged from the qualitative interviews.
Time Frame: through the completion of the study, on average 4 months.
Population: This outcome was collected aggregately to evaluate feasibility of the mobile application and to assess for generalized acceptability of the mobile application. Due to this, the results were not looked at per arm but together to assess overall qualitative themes.
Measure: Number; unit: themes
Groups:
- iCanCope + iCanCope- Contingency Management: Participants from both groups filled out qualitative survey to determine emerging themes regarding the program.
Arm/Group | iCanCope + iCanCope- Contingency Management
Number analyzed (Participants) | 82
themes
  User experience | 46
  Check-ins | 29
  Profile set up | 5
  Articles presented to the user by program | 40
  Trends presented to the user by the program | 27
  Goals presented to the user by the program | 37
  Improvement suggestions | 40
  Liked most | 36
  Liked least | 25

5. Secondary Outcome: Anxiety
Description: A comparison within change of generalized anxiety measured by the generalized anxiety disorder scale (GAD-7). After reading each statement, one of four choices are provided and respondents can select one response (1=not at all sure, 2=several days, 3=over half days, 4=nearly every day). Each column is then added, and a total score is obtained, with scores falling into four levels of anxiety, including minimal (1-4), mild (5-9), moderate (10-14), and severe (15-21)
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale
  Intake (Baseline) | 7.865 (5.21) | 7.457 (4.56) | 8.412 (6.16)
  Discharge (an average of 2 weeks) | 7.432 (5.24) | 5.667 (3.65) | 8.871 (6.48)
  Follow-Up (on average 4 months) | 6.889 (4.77) | 6.861 (4.98) | 9.697 (5.67)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P value at discharge; Test type: Superiority; p = 0.212, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; Test type: Superiority; p = 0.965, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; P value at discharge; Test type: Superiority; p = 0.294, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P value at follow-up; Test type: Superiority; p = 0.207, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; P value at follow-up; Test type: Superiority; p = 0.158, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; P value at follow-up; Test type: Superiority; p = 0.988, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

6. Secondary Outcome: Sleep Functioning
Description: A comparison within change of sleep quality measured by the PROMIS Sleep inventory. The higher the total score, the more severe the symptom. Total scores less than 24 suggest no to slight sleep disturbance, 24-28 suggest mild disturbance, 29-38 moderate disturbance, and greater than 38 severe sleep disturbance. The score has a range of 0 to 40.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 40 | 42 | 40
score on a scale | 22.4 (6.4) | 22.2 (7.3) | 21.4 (8.2)

7. Secondary Outcome: Short Form/Quality of Life
Description: the Short form survey 20- will measure quality of life across 8 subscales on respondent burden (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health). Scores were transformed linearly to 0-100 scales, with 0 and 100 assigned to the lowest and highest possible scores, where high value indicated better functioning.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale
  Intake (Baseline) | 9.342 (5.77) | 9.167 (5.02) | 10.500 (6.11)
  Discharge (an average of 2 weeks) | 9.189 (5.24) | 8.500 (4.97) | 11.206 (6.54)
  Follow-Up (on average 4 months) | 8.737 (4.84) | 9.556 (6.39) | 11.588 (6.37)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P value at discharge; Test type: Superiority; p = 0.295, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; P value at discharge; Test type: Superiority; p = 0.718, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; P value at discharge; Test type: Superiority; p = 0.738, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P value at follow-up; Test type: Superiority; p = 0.797, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; P value at follow-up; Test type: Superiority; p = 0.260, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; Test type: Superiority; p = 0.616, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

8. Secondary Outcome: Chronic Pain Acceptance
Description: Chronic Pain Acceptance Questionnaire-Revised (CPAQ-Revised) 20-item scale designed to measure acceptance of pain. The acceptance of chronic pain is thought to reduce unsuccessful attempts to avoid or control pain and thus focus on engaging in valued activities and pursuing meaningful goals will be measured across all groups. The items on the CPAQ are rated on a 7-point scale from 0 (never true) to 6 (always true). To score the CPAQ, add the items for Activity engagement and Pain willingness to obtain a score for each factor. To obtain the total score, add the scores for each factor together. Total score range is from 0 - 120, with higher scores indicating higher levels of pain acceptance.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale
  Intake (Baseline) | 65.517 (12.64) | 71.968 (11.26) | 70.148 (13.01)
  Discharge (an average of 2 weeks) | 70.606 (11.58) | 72.333 (8.26) | 67.643 (12.19)
  Follow-Up (on average 4 months) | 66.774 (9.51) | 70.462 (8.98) | 64.400 (13.30)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P value at discharge; Test type: Superiority; p = 0.333, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; P value at discharge; Test type: Superiority; p = 0.003, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; P value at discharge; Test type: Superiority; p = 0.106, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P value at follow-up; Test type: Superiority; p = 0.541, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; P value at follow-up; Test type: Superiority; p = 0.202, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; P value at follow-up; Test type: Superiority; p = 0.791, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

9. Secondary Outcome: Psychological Inflexibility in Pain Scale: Avoidance
Description: Psychological Inflexibility in Pain Scale (PIPS) Avoidance subscale is a 10-item scale used to assess psychological inflexibility in people with chronic pain will be measured across all groups. Respondents are asked to rate items on a 7-point scale that ranges from 1 (never true) to 7 (always true). The total score was calculated by summing the responses for each of the items. Higher scores indicate greater levels of psychological inflexibility. Total score range for the Avoidance subscale is 10-70. The PIPS outcome was originally registered as a single item.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale
  Intake (Baseline) | 26.361 (15.87) | 26.743 (13.28) | 25.061 (15.21)
  Discharge (an average of 2 weeks) | 22.676 (13.26) | 22.639 (11.81) | 27.194 (16.70)
  Follow-Up (on average 4 months) | 22.750 (13.56) | 22.735 (13.13) | 27.290 (14.58)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P value at discharge; Test type: Superiority; p = 0.026, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; P value at discharge; Test type: Superiority; p = 0.15, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; Test type: Superiority; p = 0.745, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P value at follow-up; Test type: Superiority; p = 0.021, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; P value at follow-up; Test type: Superiority; p = 0.155, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; P value at follow-up; Test type: Superiority; p = 0.652, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

10. Secondary Outcome: Psychological Inflexibility in Pain Scale: Cognitive
Description: Psychological Inflexibility in Pain Scale (PIPS) Cognitive subscale is a 6-item scale used to assess psychological inflexibility in people with chronic pain will be measured across all groups. Respondents are asked to rate items on a 7-point scale that ranges from 1 (never true) to 7 (always true). The total score was calculated by summing the responses for each of the items. Higher scores indicate greater levels of psychological inflexibility. Total score range for Cognitive subscale is 6-42. The PIPS outcome was originally registered as a single item.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale
  Intake (Baseline) | 23.000 (6.75) | 25.000 (6.38) | 24.324 (7.48)
  Discharge (an average of 2 weeks) | 21.833 (5.53) | 22.528 (6.58) | 23.844 (6.58)
  Follow-Up (on average 4 months) | 20.108 (6.72) | 21.800 (7.02) | 22.938 (7.50)
Statistical Analysis 1: Comparison: iCanCop+Contingency Management vs Control Group; P value at discharge; Test type: Superiority; p = 0.343, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; P value at discharge; Test type: Superiority; p = 0.995, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 3: Comparison: iCanCope vs iCanCop+Contingency Management; P value at discharge; Test type: Superiority; p = 0.371, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 4: Comparison: iCanCop+Contingency Management vs Control Group; P value at follow-up; Test type: Superiority; p = 0.228, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 5: Comparison: iCanCope vs Control Group; P value at follow-up; Test type: Superiority; p = 0.282, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 6: Comparison: iCanCope vs iCanCop+Contingency Management; Test type: Superiority; p = 0.986, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

11. Other Pre Specified Outcome: Mindfulness Based Alternative Approaches (MBAA)
Description: Do individuals with NF-1 utilize the MBAA more readily because they are on the mobile application, via Five Facet Mindfulness Questionnaire. 39-item self-completed questionnaire measuring the five facets of mindfulness: Observing (8 items), Describing (8 items), Acting with awareness (8 items), Non-judgmental (8 items), and Non-reactive (7 items). Total score ranges from 8 to 40. Higher scores indicating greater mindfulness.
Time Frame: through the completion of the study, on average 4 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | iCanCope | iCanCope+Contingency Management | Control Group
Number analyzed (Participants) | 38 | 36 | 34
score on a scale | 27.5 (3.9) | 28.2 (2.4) | 28.9 (2.5)
Statistical Analysis 1: Comparison: iCanCope+Contingency Management vs Control Group; Test type: Superiority; p = 0.421, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA
Statistical Analysis 2: Comparison: iCanCope vs Control Group; Test type: Superiority; p = 0.556, ANOVA; Reported p-values are based on Tukey's HSD post-hoc adjustment to one-way ANOVA

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | iCanCope | iCanCop+Contingency Management | Control Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT04561765/Prot_SAP_000.pdf